CLINICAL TRIAL: NCT06109012
Title: Multiple Disseminated Hydatidosis With Rare Locations: Mediastinal, Pancreatic and Pelvic: Case Report
Brief Title: Multiple Disseminated Hydatidosis With Rare Locations
Status: Completed | Type: Observational
Sponsor: Faculty Of Medicine And Pharmacy, Casablanca (Other)
Responsible Party: Principal Investigator, BENNANE WAFAA, BENNANE WAFAA, Faculty Of Medicine And Pharmacy, Casablanca
Other Study IDs: multiple hydatidose
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Echinococcus Infections
Keywords: echinococcus; serology; multiple locations
MeSH Terms: conditions — Echinococcosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: duct diversion — the patient benefited from a diversion of the bile ducts complicated by ruptured cysts with anaphylactic shock

SUMMARY:
Hydatid disease is an anthropozoonosis due to the development of the larval form of Echinococcus granulosus in the human body, which constitutes a 'dead-end' host. It's a common parasitosis in North African countries and constitutes a public health problem in Morocco. The liver and lung are the most affected while the mediastinum, pancreas and pelvis are rarely affected. We report the case of a 40-year-old patient operated 15 years ago for cerebral and cervical hydatid cysts and who was hospitalized for generalized mucocutaneous jaundice. On exploration, we discover the presence of disseminated abdominal hydatidosis with association of 3 rare locations: mediastinal, pancreatic and pelvic. Indirect diagnostic tests were positive: indirect hemagglutination (IHA) and Elisa. The Western blot test also showed the presence of specific bands, thus making it possible to retain the diagnosis of hydatidosis.

The hydatid cyst with mediastinal, pancreatic and pelvic location is rare and their association is very exceptional. It is essential to evoke the hydatid origin of any cystic lesion in a patient staying in an endemic area.

ELIGIBILITY:
Inclusion Criteria:

* none

Exclusion Criteria:

* none

Ages: 44 Years to 44 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: This is a descriptive study of a single patient with the particularity of having exceptional locations of hydatidosis.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
THE PATIENT DIED due to probably anaphylactic shock | 1 mounth
  the patient probably had the rupture of cysts during the surgical procedure with anaphylactic shock as a complication

CONTACTS AND LOCATIONS:
Locations (1):
- FMPC, Casablanca, ANFA, Morocco

IPD SHARING:
Plan to Share IPD: Undecided